CLINICAL TRIAL: NCT06376929
Title: Effect of Preoperative Low Dose Oral Carbohydrates Fluid Intake on Intraoperative Random Blood Glucose and Postoperative Nausea and Vomiting in Pediatric Patients Undergoing Ophthalmic Surgeries
Brief Title: Oral Carbohydrates in Pediatric Surgery and Random Blood Glucose Level
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Mohamed Abd El Moneim Soaida, MD, assistant professor, Cairo University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: oralcarbohydrateinpediatric
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral carbohydrate group (Active Comparator)
  Interventions: Other: oral carbohydrate containing fluid
- control group (Placebo Comparator)
  Interventions: Other: oral carbohydrate containing fluid

INTERVENTIONS:
Other: oral carbohydrate containing fluid — administration of oral carbohydrate fluid and assessment of intraoperative blood glucose level and postoperative nausea and vomiting

SUMMARY:
The correlation between preoperative oral carbohydrate intake and intraoperative random blood sugar and also the effect on postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Surgeries are considered one of the most common causes of stress response in our bodies. Common stressors include prolonged fasting, anxiety, massive tissue injury, and release of inflammatory mediators.

Hospital stay and wound healing are considered common areas of postoperative distress.

Paediatric patients undergoing surgery are subjected to stress as they are removed from their ordinary daily routine and are exposed to a number of preoperative procedures that cause anxiety and discomfort.

One major cause of discomfort and stress is the need for preoperative fasting, which is needed and accepted all over the world as a standard precaution to minimise the risk of aspiration and regurgitation during induction of general anaesthesia. Based mainly on recommendations issued by anaesthesia societies worldwide, the standard guidelines for preoperative fasting in paediatric surgery is 6 hours for solid food , 6 hours for formula milk or cow milk, 4 hours for breast milk, and 2 h for clear fluids including clear juice and water.

This strategy of preoperative fasting is a significant contributor to postoperative nausea and vomiting, other reactions such as postoperative pain , inflammatory response to surgery, and perioperative insulin resistance which is thought to affect the random blood sugar RBS. Moreover, surgical stress response causes elevation of anti insulin hormones and reduces insulin secretion which can be detrimental for surgical patients in many aspects including recovery, wound healing, and duration of hospital stay. Criticisms of standard preoperative fasting have forced practitioners to explore new ways of preparing patients for theatre. Studies previously conducted in adults exposed to cholecystectomy showed that administration of a carbohydrate beverage diminishes insulin resistance and the organs' response to trauma.

In our study we aim to address the difference between preoperative intake of oral carbohydrates and clear water on intraoperative RBS and postoperative nausea and vomiting. We thought to limit the type of surgeries to ophthalmic surgeries in an attempt to limit the discrepancy in PONV risk in different types of surgeries, higher risk of PONV and low risk of dropouts as not liable to be lengthy operations and lower risk of blood transfusion

It is thought that preoperative carbohydrate fluid intake will decrease the insulin resistance intraoperative, thus will affect the intraoperative level of random blood glucose, and post operative nausea and vomiting. This based on the idea that Preoperative fasting leads to mobilisation of lipids, increased catabolism of muscle protein, which results in ketone bodies elevation.The resulting increase in insulin resistance requires eight times the normal amount of insulin volume to maintain postoperative blood glucose at normal levels. Intraoperative catabolism is also affected by the invasiveness of the surgery, the type of anaesthesia, blood loss and body temperature, although no studies have evaluated lipid and protein catabolism but random blood glucose levels can be assessed easily and rapidly.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 3 years to 9 years
* Undergoing ophthalmic surgeries
* ASA I -II

Exclusion Criteria:

* • Parent refusal

  * Age <3 or >9
  * Underlying proemetic disease
  * Positive history of Postoperative nausea and vomiting in patient, parent or sibling
  * Currently on antiemetic medications
  * History of juvenile diabetes
  * Lengthy operations more than 3 hours
  * intraoperative Blood transfusion

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Mean values of Intraoperative random blood sugar in mg/dl | 3 months
  Mean values of Intraoperative random blood sugar in mg/dl

IPD SHARING:
Plan to Share IPD: No